CLINICAL TRIAL: NCT06073379
Title: Efficacy of Korean Manupuncture on Pain in Women With Endometriosis: a Parallel-group Randomized Controlled Trial
Acronym: ENVOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: POUHIN AOIparaM 2021
Record Dates: First submitted 2023-09-29; First posted 2023-10-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Endometriosis; Pain
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Korean manupuncture (Experimental)
  Interventions: Other: Korean manupuncture
- Placebo/control (Placebo Comparator)
  Interventions: Other: Placebo session

INTERVENTIONS:
Other: Korean manupuncture — Energy assessment on hands and body Correspondence point technique on hands Energy rebalancing with ki Maeks on hands Moxa technique on hands
  Arms: Korean manupuncture
Other: Placebo session — Energy assessment on hands and body Correspondence point technique on the hands Energy rebalancing with ki Maeks on hands (use of Qi bong) Moxa technique on hands (placebo moxas)
  Arms: Placebo/control

SUMMARY:
Endometriosis is defined as the presence and development of hormone-dependent endometrial tissue comprising both glands and stroma outside the endometrium and myometrium.

It affects 10-15% of women of childbearing age; of these, 25% are diagnosed following a consultation for infertility, and 25% following a consultation for pelvic pain.

This disease has a strong functional (pain and infertility) and organic impact, its numerous symptoms can have a considerable effect on quality of life.

Individualized analgesic management with multidisciplinary care (medical, surgical and psychological) can improve quality of life for women with endometriosis, but current treatment remains insufficient.

Korean manupuncture is a complementary treatment technique that does not interact with current treatments. It's a holistic discipline that draws up a highly detailed map of the body's correspondence on the hand. Each body zone corresponds to a zone on the hand.

The aim of this research is to evaluate the effect of Korean manupuncture on endometriosis-related pain.

Patients will be randomly assigned to 2 groups, 30 to the "Korean manupuncture" group and 30 to the "placebo/control" group. Patients will be blinded to their assigned group.

ELIGIBILITY:
Inclusion Criteria:

* Person having given oral consent
* Woman of legal age
* Woman diagnosed with endometriosis consulting for pain management

Exclusion Criteria:

* Not affiliated to the national health insurance system
* Person under legal protection (curatorship, guardianship)
* Person under court order
* Pregnant or breast-feeding women
* Menopausal women (menopause is defined as amenorrhea lasting more than 12 consecutive months)
* An adult unable to give consent
* Women who have had a hysterectomy
* Women who cannot speak or read French
* Hands not accessible for treatment
* Inability to follow the entire protocol
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Variation in the Visual Analog Scale (VAS) | Between Day 1 and Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France